CLINICAL TRIAL: NCT04852367
Title: PanDox: Feasibility of Enhanced Chemotherapy Delivery to Non-resectable Primary Pancreatic Tumours Using Thermosensitive Liposomal Doxorubicin (ThermoDox®) and Focused Ultrasound
Brief Title: PanDox: Targeted Doxorubicin in Pancreatic Tumours
Acronym: PanDox
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Imunon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OCTO_095
Record Dates: First submitted 2021-04-07; First posted 2021-04-21 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer Stage IV; Pancreatic Cancer Non-resectable; Pancreatic Cancer Metastatic
Keywords: Focused ultrasound; Doxorubicin; Thermodox; Thermosensitive Liposome; Drug delivery
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Doxorubicin

STUDY DESIGN:
Intervention Model Description: prospective non-randomised safety cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Doxorubicin) (Active Comparator): a single intravenous dose of Doxorubicin, 50 mg/ m2 in 250 mL of normal saline or 5% dextrose over a 30-min infusion is delivered as per local practice.
  Interventions: Drug: Doxorubicin
- Arm B (ThermoDox + Focused Ultrasound) (Experimental): under general anaesthetic, patients receive FUS, which is moved through the target tumour volume to raise the bulk tumour temperature above the thermal release threshold. At presumed target temperature, a single intravenous dose of ThermoDox®, 50 mg/ m2 in 250 mL of normal saline or 5% dextrose over a 30-min infusion is delivered concurrently to FUS, in line with the pharmacy manual provided by the manufacturer. FUS will continue following infusion, for no longer than two hours from infusion commencing.
  Interventions: Device: Focused Ultrasound; Drug: ThermoDox

INTERVENTIONS:
Device: Focused Ultrasound — Focused ultrasound targetting the tumour at subablative powers, to facilitate drug release
  Arms: Arm B (ThermoDox + Focused Ultrasound)
Drug: Doxorubicin — Doxorubicin infusion
  Arms: Arm A (Doxorubicin)
Drug: ThermoDox — ThermoDox infusion
  Arms: Arm B (ThermoDox + Focused Ultrasound)

SUMMARY:
This study will combine focused ultrasound to generate heat, and a heat-sensitive chemotherapy drug (ThermoDox®), delivered into the blood of participants with non-resectable pancreatic cancer. We will compare this to standard delivery of chemotherapy - the drug Doxorubicin given into the blood without the addition of ultrasound. We aim to determine whether the novel approach to delivering chemotherapy with heating the tumour by focused ultrasound can enhance the amount of drug delivered to pancreatic tumours. This will be measured by analysing a biopsy sample of treated tumour.

DETAILED DESCRIPTION:
PanDox is a phase I prospective, non-randomised, safety cohort study with the primary aim to quantify the enhancement in delivery of intratumoural doxorubicin concentration in pancreatic tumours, for a given systemic dose. Drug release is triggered from systemically circulating ThermoDox® by highly localized hyperthermia induced by extracorporeal ultrasound-guided FUS device at sub-ablative powers.

The study will have all patients recruited from a single UK site (Oxford) and will comprise adult patients with non-resectable pancreatic adenocarcinomas.

Patients referred to Oncology will have cross-sectional imaging reviewed for suitability of tumour targeting, and MDT (Multi-Disciplinary Team) agreement before being approached. Screening comprises clinical history and examination, routine blood tests, cardiac assessment by ECG (Electrocardiogram) and ECHO (Echocardiogram), abdominal ultrasound examination and a pre-operative assessment to ensure suitability for general anaesthetic. Suitability of potential target lesions will be based on ultrasound examination.

The study has an open label design with all participants receiving a single dose of either standard doxorubicin OR systemic ThermoDox® with ultrasound guided FUS targeted at a pancreas tumour using the Model JC200 Focused Ultrasound Tumour Therapeutic System (Haifu Medical, JC200), which is clinically approved (CE-marked) for tumour therapy in Europe and China.

Participants who successfully complete screening will be allocated to either Arm A (doxorubicin) or Arm B (ThermoDox® with FUS) based on pre-determined checklist. This is to ensure feasibility and safety of patients to undergo FUS. It also permits patients who have successfully completed screening, but who are not suitable for FUS, to participate in a clinical trial.

Baseline imaging is performed in the week prior to intervention and consists of fluorodeoxyglucose (18F-FDG) positron emission tomography / CT (PET-CT) for all patients. Participants in Arm B also undergo dynamic contrast-enhanced Magnetic Resonance Imaging (DCE-MRI).

For Arm A patients: following pre-medications, a single intravenous dose of Doxorubicin, 50 mg/ m2 in 250 mL of normal saline or 5% dextrose over a 30-min infusion is delivered as per local practice.

For Arm B patients: a single pancreatic tumour (or partial tumour volume), is targeted for drug delivery.

Patients will receive pre-medications and general anaesthetic (Fig. 1b), In order to minimise respiratory movement of the target tumour during the intervention, appropriate anaesthetic techniques, such as high-frequency jet ventilation may be employed. High intensity focused ultrasound to cause a small area of tumour ablation will be used to help confirm location targeting accuracy and may give a treatment reference point for Endoscopic Ultrasound Sampling (EUS) biopsy. No more than 2 ablation spots will be applied. Once confirmed, lower-intensity FUS is then moved through the target tumour volume to raise the bulk tumour temperature above the thermal release threshold. This is based on an individualised plan of FUS parameters (power, duty cycle, scanning speed, unit spacing), devised from patient imaging and computer modelling, accounting for differences in propagation path length and overlying tissue structures. (Gray et al., 2019) At target temperature, a single intravenous dose of ThermoDox®, 50 mg/ m2 in 250 mL of normal saline or 5% dextrose over a 30-min infusion is delivered concurrently to FUS, in line with the pharmacy manual provided by the manufacturer. FUS will continue following infusion, for no longer than two hours from infusion commencing.

FUS-mediated hyperthermia is delivered under ultrasound guidance using clinically approved treatment modes of the therapeutic device, namely either linear (moving beam) or dot (shot-by-shot) mode, using the on-board plane-by-plane treatment planning tool to encompass all or part of the target tumour volume. Device settings are chosen to achieve hyperthermia in the range of 40-42 °C in the target region. The specific treatment parameters will naturally vary depending on tumour anatomy The addition of a passive material layer for beam expansion may be used to expand the beam size for optimal heating control and efficiency. Supplemental hand-held diagnostic ultrasound probes may be used during treatment to monitor and quantify natural target motion and/or the presence of cavitation.

For all patients, tumour sampling for primary end point will be acquired via EUS, performed within thirty hours of treatment. These will be analysed using a Good Laboratory Practice-validated high performance liquid chromatography (HPLC) assay, to quantify doxorubicin at the targeted site. Plasma samples are collected immediately before the start of ThermoDox® infusion, immediately after completion of ThermoDox® infusion, and immediately after completion of FUS exposure, to evaluate doxorubicin pharmacokinetics.

In the post-treatment period, Arm B patients will have a repeat DCE-MRI scan for comparison with baseline. Additionally, all study patients will have follow-up imaging performed at 21days following intervention to assess potential response in the target tumour activity and volume.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent prior to any screening procedures being performed and is able and willing to comply with the protocol and its requirements.
* Male or Female, aged 18 years or above.
* Prior histological confirmation of pancreatic adenocarcinoma

  * Non-resectable or metastatic (stage IV)
  * The primary pancreatic lesion measuring at least 1.5cm minimum diameter and amenable to EUS biopsy sampling
* ECOG performance status 0-1 (Appendix 1)
* Left ventricular ejection fraction (LVEF) ≥ 50% as determined by echocardiogram
* Willing to allow his or her General Practitioner and Consultant, if appropriate, to be notified of participation in the trial.
* Life expectancy of at least 3 months
* Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use highly effective contraception during the trial and for 6 months thereafter.
* Participant has clinically acceptable laboratory results during screening window:

Lab Test Value required Haemoglobin (Hb) (transfusion to achieve this allowed) ≥ 9g/dL Neutrophils ≥ 1.5 109/L Platelet count ≥ 100 109/L ALT ≤ 2.5 x ULN Alkaline phosphatase ≤ 5 x ULN Serum Bilirubin (stenting to achieve this allowed) ≤ 1.5 x ULN Creatinine Clearance (Calculated by Cockcroft-Gault criteria) ≥ 50ml/min INR <1.5 unless taking oral anticoagulant (this to be stopped at least 1 week prior to biopsy, at which point this INR limit will then apply)

Exclusion Criteria:

A patient will be ineligible for inclusion in this study if any of the following criteria apply:

* Significant renal or hepatic impairment.
* Unstable ischemic heart disease, cardiac dysrhythmias, coronary/peripheral artery bypass graft or cerebrovascular accident within 6 months prior to starting treatment
* Uncontrolled arterial hypertension despite medical treatment.
* Ongoing congestive heart failure or cardiac dysrhythmias of NCI CTCAE Grade ≥2 or uncontrolled atrial fibrillation.
* On-going significant infection (chest, urine, blood, intra-abdominal).
* Uncontrolled diabetes.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such procedure
* Previous targeted therapies to the pancreatic adenocarcinoma (including radiofrequency ablation or radiotherapy)
* History of other malignancy less than 3 years before the diagnosis of current cancer, EXCLUDING the following: Non-melanoma skin cancer, in situ carcinoma of the cervix treated surgically with curative intent, other malignant tumours that have been treated curatively and patient is deemed disease-free
* Endocrine therapy - patients with prostate cancer may continue to receive endocrine therapy to maintain castrate levels of androgens
* Known allergic reactions to any of the drugs or liposomal components or intravenous imaging agents used in this study
* Resting ECG with QTc >480msec at 2 or more time points within a 24h period (using Fredericia correction).
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that the investigator considers would make the patient a poor trial candidate, would impart excess risk associated with study participation or drug administration or could interfere with protocol compliance or the interpretation of trial results.
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial. However, those female patients who have a negative serum pregnancy test before enrolment and agree to use one highly effective form of contraception (oral, injected or implanted hormonal contraception or intrauterine device) in addition to condom plus spermicide, for four weeks before entering the trial, during the trial and for six months afterwards are considered eligible.
* Male patients with partners of child-bearing potential unless they agree to take measures not to father children by using one form of highly effective contraception including: oral, injected or implanted hormonal contraception or intra-uterine device in addition to condom plus spermicide, during the trial and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (condom plus spermicidal gel) during the trial and for six months afterwards to prevent exposure to the foetus or neonate.
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.
* Severe immunologic defect or compromised bone marrow function.
* Patients who are serologically positive for Hepatitis B, Hepatitis C or HIV.
* Previous doxorubicin and epirubicin must not have exceeded 450 mg/m2 and 900 mg/m2, respectively.
* Patients who have a contraindication to MRI scans, for example patients who have a cardiac pacemaker, will be excluded from Arm B (as per Arm Assignment criteria, Appendix 3 of protocol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
To quantify the enhancement in intratumoural doxorubicin concentration when delivered with ThermoDox® and mild hyperthermia generated non-invasively by focused ultrasound (FUS) compared to free drug alone | within 30 hours of intervention
  A statistically significant enhancement in concentration of total intra-tumoural doxorubicin from tumour biopsies at the targeted tumour site receiving drug with FUS compared to drug alone. Quantification of inter-tumoural drug release will be achieved using a GLP HPLC (High Pressure Liquid Chromatography) assay

SECONDARY OUTCOMES:
Number of adverse events related to ThermoDox® and FUS compared to free drug alone | for 21 days post intervention
  No statistically significant increase in low grade (I-II) adverse events related to drug+FUS cf drug alone, according to toxicities graded by NCI CTCAE v5.0
  No statistically significant increase in high grade (III and above) adverse events related to drug+FUS cf drug alone, according to toxicities graded by NCI CTCAE v5.0
Change in radiologically-assessed tumour activity in patients treated with ThermoDox® and FUS, compared to free drug alone | Pre-treatment, and 14 days post treatment
  A statistically significant reduction in tumour activity between targeted tumour sites receiving drug with FUS, compared to drug alone, as determined either by SUVmax or by PERCIST response criteria (SULpeak) on FDG-PET-CT scans performed pre- and post intervention.
Change in patient symptom scores in patients with pancreatic cancer treated with of ThermoDox® and FUS compared to those treated with doxorubicin | Pre-treatment, within 30 hours post treatment, 14 days and 21 days post treatment
  No significant difference in patient symptom scores following treatment with FUS with ThermoDox® vs Doxorubicin alone, according to a pancreatic cancer-specific Quality of Life questionnaire (EORTC QLQ - PAN26)

OTHER OUTCOMES:
To assess effects of ThermoDox® and FUS treatment compared to free drug alone on pancreatic tumour biomarkers | Taken pre-treatment and 21 days post-treatment
  A statistically significant reduction in tumour markers CA19-9 and CEA as measured pre and post treatment, in plasma samples

CONTACTS AND LOCATIONS:
Overall Officials: Mark Middleton, Principal Investigator — Consultant Medical Oncologist and Professor of Experimental Cancer Medicine
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Plan to anonymise patient data (assigned trial number) and results to be published in peer reviewed journal as anonymous data points/averaged data

REFERENCES:
- [Derived] Spiers L, Gray M, Lyon P, Sivakumar S, Bekkali N, Scott S, Collins L, Carlisle R, Wu F, Middleton M, Coussios C. Clinical trial protocol for PanDox: a phase I study of targeted chemotherapy delivery to non-resectable primary pancreatic tumours using thermosensitive liposomal doxorubicin (ThermoDox(R)) and focused ultrasound. BMC Cancer. 2023 Sep 23;23(1):896. doi: 10.1186/s12885-023-11228-z. PMID 37741968